CLINICAL TRIAL: NCT04369404
Title: Impact of Decision Aids in Urogynecology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director, Health Decision Sciences Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017P001883 - 01
Record Dates: First submitted 2020-03-24; First posted 2020-04-30 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence; Overactive Bladder
Keywords: shared decision making
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: A usual care arm was recruited first, then the intervention arm was recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): In the usual care group, the providers do not have access to the decision aids.
- Patient Decision Aid (Experimental): Providers have access to patient decision aids to review and discuss during the visit.
  Interventions: Behavioral: Pelvic organ prolapse decision aid; Behavioral: Stress urinary incontinence decision aid; Behavioral: Overactive bladder decision aid

INTERVENTIONS:
Behavioral: Pelvic organ prolapse decision aid — Paper-based educational tool to guide shared decision making conversations for treatment of pelvic organ prolapse
  Arms: Patient Decision Aid
Behavioral: Stress urinary incontinence decision aid — Paper-based educational tool to guide shared decision making conversations for treatment of stress urinary incontinence.
  Arms: Patient Decision Aid
Behavioral: Overactive bladder decision aid — Paper-based educational tool to guide shared decision making conversations for treatment of overactive bladder.
  Arms: Patient Decision Aid

SUMMARY:
To evaluate how patient knowledge and confidence in decision making can be impacted by shared decision making in common urogynecology conditions.

DETAILED DESCRIPTION:
The investigators will enroll patients seeing a specialist to discuss treatment of pelvic organ prolapse, overactive bladder and stress urinary incontinence in this pilot study. The study will evaluate the feasibility and acceptability of three decision aids designed to promote shared decision making conversations for these three condition. The investigators use a quasi-experimental design in which the investigators first enroll patients in the control arm and measure their outcomes. Then, the investigators enroll patients into the intervention arm and measure their outcomes. The investigators estimate that it will take about one month to recruit the control arm and one month to recruit the intervention arm. Patients will be surveyed after the clinic visit with a specialist and surveys will assess patients' knowledge, treatment preferences, shared decision making, decisional conflict and acceptability of the tool. A clinician survey will be administered and completed after each patient visit, that details how the physician felt about the length of the visit, how informed the patient was, and how far along they may be with their decision.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-95 years only
* English speaking
* Pelvic organ prolapse defined by noticeable (to the patient) vaginal bulging
* Symptoms of stress urinary incontinence (cough, sneeze, laugh, exercise)
* Presenting for initial consultation for either of the above symptoms

Exclusion Criteria:

* Primary complaint is not vaginal bulging or stress urinary incontinence
* Prior surgery for pelvic organ prolapse or any incontinence procedure

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Recruiting only female patients as Urogynecology conditions only affect women's pelvic organs and pelvic floor.
Enrollment: 66 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques F, Josloff K, Hung K, Wakamatsu M, Sepucha KR. Decision aids and shared decision making in urogynecology. Menopause. 2021 Dec 13;29(2):178-183. doi: 10.1097/GME.0000000000001901. PMID 34905749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were patients who had scheduled a visit with the Female Pelvic Medicine and Reconstructive Surgery Division of the Obstetrics and Gynecology Department at Massachusetts General Hospital between February 2019 - April 2019
  Eligible patients were English speaking and between 18-95 years old. They had scheduled a visit for either pelvic organ prolapse, stress urinary incontinence, or overactive bladder.
Pre-assignment Details: Patients with prior surgery for pelvic organ prolapse or incontinence, or did not attend the scheduled visit were ineligible.
Period: Overall Study
Arm/Group | Usual Care | Patient Decision Aid
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Patient Decision Aid | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.7) | 60.2 (14.6) | 58.9 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants] — Participants were recruited from the Urogynecology Clinic at the Massachusetts General Hospital in Boston, MA
  participants
    United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Patient Knowledge
Description: Patients completed four multiple choice knowledge items for each condition and a total knowledge score (0-4) was calculated. The score was converted to a 0-100% scale, with higher scores indicating higher knowledge.
Time Frame: Within 1 day
Population: Anyone who answered the knowledge items.
Measure: Mean (Standard Deviation); unit: percentage of questions answered correct
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
percentage of questions answered correct | 60 (30) | 72 (21)
Statistical Analysis 1: Comparison: Usual Care vs Patient Decision Aid; Test type: Superiority — We hypothesize that participants who received the decision aid will have higher knowledge. This is pilot study, thus we did not have a power calculation; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 12, 95% CI 2-sided [0.7 to 24.6]

2. Primary Outcome: Patient Treatment Preference
Description: 1 item assess patients' preferred treatment- Response options included no treatment at this time, conservative and non conservative options, or I am not sure. Responses were categorized into clear treatment preference (no treatment, conservative and non-conservative options) vs unsure (I am not sure) treatment preference.
Time Frame: Within 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
Participants
  clear treatment preference | 22 | 28
  unsure treatment preference | 11 | 5
Statistical Analysis 1: Comparison: Usual Care vs Patient Decision Aid; a chisquare test was conducted to determine if the proportion of treatment "unsure" responses were different between the usual care and intervention arms; Test type: Other; p = 0.085, Chi-squared; Pearson Chi-Square = 2.970

3. Primary Outcome: Physician Visit Satisfaction
Description: Physicians answered 1 item on how satisfied they were with the visit: Extremely satisfied, Very satisfied, Somewhat satisfied, and Not at all satisfied
Time Frame: Within 1 day
Population: Physicians were not considered enrolled in the study, but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
Participants
  Not at all satisfied | 0 | 0
  Somewhat satisfied | 5 | 9
  Very satisfied | 23 | 19
  Extremely satisfied | 5 | 5
Statistical Analysis 1: Comparison: Usual Care vs Patient Decision Aid; Test type: Other; p = 0.47, Chi-squared; Pearson Chi-Square = 1.524

4. Secondary Outcome: SURE Scale
Description: Measures decisional conflict, consists of 4 yes/no items. Total scores range 0-4 where 4 indicates no decisional conflict and scores less than or equal to 3 indicate decisional conflict. The number of participants who got a total score of 4, indicating no decisional conflict, is reported
Time Frame: Within 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
Participants | 24 | 30

5. Secondary Outcome: CollaboRATE
Description: Three items ask patients to rate their provider on a scale of 1-10, with 10 being outstanding. The measure is a dichotomized score. Participants who reported a "10" on all 3 items were "topscored" into one group; everyone else were categorized into another group. The number of participants who gave a topscore (a "10" for all 3 items) was reported.
Time Frame: Within 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
Participants | 17 | 25

6. Secondary Outcome: SDM Process Scale
Description: Four items that measures the amount of shared decision making that occurs in an interaction. Total scores ranged from 0-4, with higher scores indicating more shared decision making occurred.
Time Frame: Within 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
score on a scale | 3.18 (0.88) | 3.17 (0.85)

7. Secondary Outcome: MD Perceptions of Length of Visit
Description: One item assessed how physician felt about the length of the visit. Responses were: Shorter than normal, About normal, Longer than normal. Number of physicians who responded that the visit was "shorter than normal" or "about normal" is reported.
Time Frame: Within 1 day
Population: Physicians were not considered enrolled in the study, but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patient Decision Aid
Number analyzed (Participants) | 33 | 33
Participants | 25 | 23

ADVERSE EVENTS:
Time Frame: Participants were assessed within one day of survey receipt. The surveys were completed within 2 weeks of the visit and were checked as they came in for evidence of adverse events.
Arm/Group | Usual Care | Patient Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04369404/Prot_SAP_000.pdf